CLINICAL TRIAL: NCT03071900
Title: Enumeration and Molecular Characterization of Circulating Tumor Cells (CTCs) Using a in Vivo Device in Squamous Cell Carcinoma of Head and Neck (SCCHN)
Brief Title: CTC Detection Rate in SCCHN With a in Vivo Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NJTRH_CellColletor01
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Circulating Tumor Cell; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Neoplastic Cells, Circulating; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCCHN (Experimental): squamous cell carcinoma of the head and neck
  Interventions: Diagnostic Test: circulating tumor cell analysis
- Control (Experimental): health volunteers
  Interventions: Diagnostic Test: circulating tumor cell analysis

INTERVENTIONS:
Diagnostic Test: circulating tumor cell analysis — Detect circulating tumor cells with CellCollector in SCCHN and control group.

SUMMARY:
Detection rate and isolation yield of CTC is low in squamous cell carcinoma of head and neck (SCCHN) with in vitro approaches rely on limited sample volumes. In this study, we applied a new method, the CellCollector, which could capture CTC in vivo from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* SCCHN confirmed with clinical examination
* Have agreed to undergo CTC analysis in vivo;
* ECOG：0-2

Exclusion Criteria:

* the other cancer types

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-03-15 (Estimated); Study Completion 2017-04-20 (Estimated)

PRIMARY OUTCOMES:
CTC isolation | 9 month
  Isolate circulating tumor cells in vivo with CellCollector

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Tongren Hospital, Nanjing, Jiangsu, China